CLINICAL TRIAL: NCT04830592
Title: A Multicentre, Open-label, Dose-escalating, Phase Ib, Study of Intravenous Dosing of NG-641, as Monotherapy or in Combination With Pembrolizumab in Patients With Surgically Resectable Squamous Cell Carcinoma of the Head and Neck
Brief Title: A Study of NG-641 and Pembrolizumab in Squamous Cell Carcinoma of the Head and Neck
Acronym: MOAT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Akamis Bio (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NG-641-02
Record Dates: First submitted 2021-03-31; First posted 2021-04-05 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2024-08

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
Keywords: Squamous cell carcinoma of the head and neck; SCCHN; NG-641; Pembrolizumab; Akamis Bio
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Part A (Experimental): NG-641 monotherapy
  Interventions: Biological: NG-641
- Part B (Experimental): NG-641 and pembrolizumab
  Interventions: Biological: NG-641; Biological: Pembrolizumab

INTERVENTIONS:
Biological: NG-641 — Patients receive three doses of NG-641 by intravenous infusion. NG-641 is a replication competent adenoviral vector producing a bispecific T cell activator (TAc) targeting fibroblast activation protein (FAP) plus immune enhancer genes CXCL9/CXCL10/IFNa2. This can lead to killing of tumor cells and stimulation of immunity against the tumor cells.
Biological: Pembrolizumab — Patients receive three doses of NG-641 by intravenous infusion and a single dose of Pembrolizumab by intravenous infusion.
  Arms: Part B

SUMMARY:
A multicentre, open-label, non-randomized, phase Ib neoadjuvant study of intravenous NG-641, as monotherapy or in combination with pembrolizumab, in patients with surgically resectable squamous cell carcinoma of the head and neck (SCCHN).

DETAILED DESCRIPTION:
Part A (NG-641 monotherapy): Approximately 16 evaluable patients will receive three doses of IV NG-641 in Part A. Patients will then proceed to planned surgical resection.

Part B (NG-641 and pembrolizumab): Up to 20 evaluable patients will receive three doses of IV NG-641 and one dose of pembrolizumab. Patients will then proceed to planned surgical resection.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed or recurrence of clinical stage III-IVb, histologically confirmed oral cavity, larynx, hypopharynx or oropharynx SCCHN (T1 with N2-3; T2 with N2-3; T3 with N0-3; T4a with N0-3)
2. Disease is considered resectable, definitive surgery is planned in the next 8 weeks from screening, and the patient is willing to undergo surgery (potential for 2-3 cm of resected tumour specimen to be available for translational research purposes)
3. Provide written informed consent to participate
4. Aged 18 years or over
5. Willing to consent to tumour biopsies at baseline
6. ECOG performance status 0 or 1
7. Ability to comply with study procedures in the Investigator's opinion
8. Adequate renal function
9. Adequate hepatic function
10. Adequate bone marrow function
11. Meeting reproductive status requirements

Exclusion Criteria:

1. Prior allogeneic or autologous bone marrow or organ transplantation
2. Active infections requiring antibiotics, physician monitoring or recurrent fevers (>38.0˚C) associated with a clinical diagnosis of active infection. Active infection requiring systemic therapy within 1 week of the anticipated first dose of study drug
3. Active viral disease or positive test for hepatitis B virus, hepatitis C virus (HCV) or HIV/AIDS
4. Patients who have active autoimmune disease that has required systemic therapy in the past 2 years, are immunocompromised in the opinion of the Investigator, or are receiving systemic immunosuppressive treatment (see protocol for full criteria)
5. Treatment with any COVID-19 vaccine in the 28 days before the first dose of NG-641, unless the vaccine is known to not be based on an adenoviral vector (e.g., mRNA vaccines)
6. Treatment with any vaccine (including known non-adenoviral COVID-19 vaccines) in the 7 days before first dose of NG-641
7. History of clinically significant chronic liver disease
8. History of clinically significant interstitial lung disease (including pneumonitis)
9. History of prior Grade 3-4 acute kidney injury or other clinically significant renal impairment
10. Use of antiviral agents
11. Incomplete recovery from surgery, incomplete healing of an incision site or evidence of infection
12. Any of the following in the 3 months before the first dose of study treatment: Grade 3 or 4 gastrointestinal bleeding or risk factors for gastrointestinal bleeding, infectious or inflammatory bowel disease, pulmonary embolism or other uncontrolled thromboembolic event, history or evidence of haemoptysis, or significant cardiovascular or cerebrovascular event
13. Any known Common Terminology Criteria for Adverse Events (CTCAE) Grade ≥2 coagulation abnormality/coagulopathy
14. Prior history of bowel obstruction, or infectious or inflammatory bowel disease in the 3 months before the first dose of study treatment
15. Major surgery or treatment with any chemotherapy, radiation therapy, biologics for cancer or investigational drug/therapy in the 28 days before the first dose of study treatment:

    • All toxicities attributed to prior anti-cancer therapy other than alopecia must have resolved to Grade 1 or baseline before the first dose of study treatment. Patients with toxicities (other than renal toxicities) attributed to prior anti-cancer therapy which are not expected to resolve and result in long lasting sequelae, such as neuropathy after platinum-based therapy, are permitted to enrol
16. Other prior malignancy active within the previous 3 years
17. Tumour location/extent considered by the Investigator to present a significant risk of airway obstruction if tumour flare or necrosis were to occur
18. Any serious or uncontrolled medical disorder that, in the opinion of the Investigator or the Medical Monitor, may increase the risk associated with study participation or study treatment administration, impair the ability of the patient to receive protocol therapy or interfere with the interpretation of study results
19. Previous treatment with any other enadenotucirev-based therapy, or fibroblast activation protein (FAP) targeting agent
20. Known allergy/immune-related adverse reactions to NG-641 transgene or immune checkpoint inhibitor products or formulation; severe hypersensitivity to another monoclonal antibody
21. Any other medical or psychological condition that would affect the patient's ability to comply with all visits and assessments, or compromise ability to give informed consent
22. Related to or a dependent of the site staff, or a member of the site staff.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-11-04 (Actual); Primary Completion 2023-12-07 (Actual); Study Completion 2024-10-04 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (safety and tolerability) | End of Study Treatment Visit (Day 57)
  Assess the safety and tolerability of NG-641 by review of adverse events (AEs), serious adverse events, AEs resulting in delays to planned surgery, AEs leading to study treatment or study discontinuation and AEs resulting in death.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Ottensmeier, Prof., Principal Investigator — The Clatterbridge Cancer Centre
Locations (4):
- United Kingdom (4):
  - Cardiff & Vale University LHB, Cardiff
  - The Clatterbridge Cancer Centre, Liverpool
  - The Royal Marsden Hospital, London
  - University Hospital Southampton NHS Foundation Trust, Southampton

REFERENCES:
- [Derived] Khalil DN, Prieto Gonzalez-Albo I, Rosen L, Lillie T, Stacey A, Parfitt L, Soff GA. A tumor-selective adenoviral vector platform induces transient antiphospholipid antibodies, without increased risk of thrombosis, in phase 1 clinical studies. Invest New Drugs. 2023 Apr;41(2):317-323. doi: 10.1007/s10637-023-01345-8. Epub 2023 Mar 10. PMID 36897458